CLINICAL TRIAL: NCT03429595
Title: Randomized, Double-Blind, Vehicle Controlled, Phase 2 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Activity of Topical ATx201 GEL (2% and 4%) in Outpatients With Impetigo
Brief Title: Study Evaluating the Safety, Tolerability, PK, and Activity of Topical ATx201 Gel in Outpatients With Impetigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATx201-004
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned (stratified by age) by using an Interactive Web Response System (IWRS) to one of five treatment groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: ATx201 GEL 2% (Experimental)
  Interventions: Drug: ATx201
- Group 2: ATx201 GEL 4% (Experimental)
  Interventions: Drug: ATx201
- Group 3: ATx201 GEL 4% plus vehicle (Experimental)
  Interventions: Drug: ATx201; Other: ATx201 GEL Vehicle
- Group 4: ATx201 GEL 4% plus vehicle (Experimental)
  Interventions: Drug: ATx201; Other: ATx201 GEL Vehicle
- Group 5: Vehicle (Placebo Comparator)
  Interventions: Other: ATx201 GEL Vehicle

INTERVENTIONS:
Drug: ATx201 — ATx201 GEL
  Arms: Group 1: ATx201 GEL 2%; Group 2: ATx201 GEL 4%; Group 3: ATx201 GEL 4% plus vehicle; Group 4: ATx201 GEL 4% plus vehicle
Other: ATx201 GEL Vehicle — Vehicle
  Arms: Group 3: ATx201 GEL 4% plus vehicle; Group 4: ATx201 GEL 4% plus vehicle; Group 5: Vehicle

SUMMARY:
This is a Phase 2 study evaluating the safety, tolerability, systemic exposure, and activity of topical ATx201 GEL (2% and 4%) treatment for 1, 2, or 5 days in outpatients with primary nonbullous or bullous impetigo.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary nonbullous or bullous impetigo
* affected area comprising 1 to 100 cm2 with surrounding erythema not extending more than 2 cm from the edge of any affected area.
* target area has total SIRS score of at least 3, including pus/exudate of at least 1
* normally active and otherwise in good health by medical history and physical examination

Exclusion Criteria:

* has a pre-existing skin condition or skin trauma with clinical evidence of secondary infection
* has an infection that could not be appropriately treated with a topical antibiotic or severe manifestation of impetigo warranting systemic therapy
* clinically significant mental illness
* pregnant or breast-feeding
* recent history, or strong potential for, alcohol or substance abuse.
* skin condition that may interfere with the placement of study treatment or impede clinical evaluations
* receipt of systemic drugs that affect the immune system within the past 3 months
* receipt of any topical medication on the regions to be treated or topical antibiotics used for nasal decolonization within the past 24 hours

Ages: 9 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Incidences of Adverse Events and Laboratory Parameters | 14 days
  incidences of adverse events reports and changes in significant laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Director — CMO
Locations (16):
- South Africa (16):
  - AntibioTx Investigational Site, Bloemfontein
  - AntibioTx Investigative Site, Boksburg
  - AntibioTx Investigative Site, Claremont
  - AntibioTx Investigative Site, Durban
  - AntibioTx Investigative Site, eMkhomazi
  - AntibioTx Investigative Site, Germiston
  - AntibioTx Investigative Site 2, Johannesburg
  - AntibioTx Investigative Site, Johannesburg
  - AntibioTx Investigative Site, Kraaifontein
  - AntibioTx Investigative Site, Mpumalanga
  - AntibioTx Investigative Site, Paarl
  - AntibioTx Investigative Site 2, Port Elizabeth
  - AntibioTx Investigative Site, Port Elizabeth
  - AntibioTx Investigative Site, Pretoria
  - AntibioTx Investigative Site, Soshanguve
  - AntibioTx Investigative Site, Winnie Mandela

IPD SHARING:
Plan to Share IPD: No